CLINICAL TRIAL: NCT01085383
Title: Aripiprazole Treatment for Antipsychotic Induced Hyperprolactinaemia in Patients With Severe Mental Illness and Learning Disabilities
Brief Title: Aripiprazole and Prolactin Study
Acronym: APS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCTUMI-03; 2009-011228-73 (EudraCT Number)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Hyperprolactinemia
Keywords: Antipsychotic; hyperprolactinemia; hypogonadism; aripiprazole
MeSH Terms: conditions — Hyperprolactinemia; Hypogonadism | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole will be started at 5 mg daily and increased in a treat-to-target fashion by 5 mg steps until the primary outcome or the maximum tolerated or permitted dose of 30 mg is reached
  Other Names: Abilify

SUMMARY:
Antipsychotic medicines are used routinely in people with severe mental illness or learning disability. Antipsychotics often induce hyperprolactinemia (high prolactin level) and in almost all women, and some men, this causes hypogonadism (impaired ovarian or testicular function)often with osteoporosis, partly explaining psychiatric patients' high fracture risk. Reducing prolactin by changing antipsychotic or adding a dopamine agonist often worsens psychosis. Adding aripiprazole to current antipsychotic normalizes prolactin in adult schizophrenic patients, without serious side effects. We thus plan a study of add-on aripiprazole in people with antipsychotic induced hyperprolactinemia.

Our main hypothesis is that aripiprazole will normalize or reduce prolactin sufficiently to restore normal ovarian and testicular function. Our secondary hypothesis is that restoration of normal ovarian and testicular function will improve bone mineral density in patients in whom this was reduced at the time of entry into the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to give informed consent for participation in the study.
* Males or Females, aged 16-50 years (women), 16-60 (men).
* Diagnosed with antipsychotic induced hyperprolactinaemia of sufficient severity to induce secondary hypogonadism.
* Stable dose of current regular antipsychotic medication for at least three months prior to study entry.
* Female participants of child bearing potential willing to ensure that they or their partner use effective contraception during the study and for 1 month thereafter
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant to be notified of participation in the study.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Plans to donate blood during the study
* Participants who have participated in another research study involving an investigational product in the past 8 weeks
* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Plans to donate blood during the study
* Participants who have participated in another research study involving an investigational product in the past 8 weeks

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Normalization or reduction in prolactin sufficient to restore gonadal function | Monthly and then 6 monthly intervals over 2 years
  Prolactin and sex hormones will be measured on addition of aripiprazole to current antipsychotic treatment. Aripiprazole will be started at 5 mg and uptitrated in a treat-to-target fashion by 5 mg at monthly intervals until prolactin has normalized or decreased sufficiently to restore menses in the women and a normal testosterone in the men. Maximum aripiprazole dose will be 30 mg.

SECONDARY OUTCOMES:
Normalization or improvement in bone mineral density | 2 years
  Bone mineral density will be measured at baseline in patients aged 20 years or older with a presumed duration of hypogonadism of minimum one year. The measurement will be repeated in those with a low bone mineral density at baseline after two years aripiprazole treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guy M Goodwin, PhD, Principal Investigator — University of Oxford
Locations (1):
- University Dept. of Psychiatry, Oxford, Oxfordshire, United Kingdom